CLINICAL TRIAL: NCT05896527
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Dose-ranging Study to Evaluate the Efficacy and Safety of DC-806 in Participants With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of DC-806 in Participants With Moderate to Severe Plaque Psoriasis
Acronym: Illuminate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCE806201; 2022-502249-90-00 (Other: EU CTR Number); J5B-MC-FHAG (Other: DICE Therapeutics, a wholly owned subsidiary of Eli Lilly and Company)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The Sponsor, participants, Investigators, and study staff responsible for any study procedures was blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo tablets orally twice daily (BID) for 12 weeks.
  Interventions: Other: Placebo
- DC-806 200 mg BID (Experimental): Participants received 200 milligrams (mg) of DC-806 tablets orally twice daily for 12 weeks.
  Interventions: Drug: DC-806
- DC-806 400 mg BID (Experimental): Participants received 400 mg of DC-806 tablets orally twice daily for 12 weeks.
  Interventions: Drug: DC-806
- DC-806 600 mg QD (Experimental): Participants received 600 mg of DC-806 tablets orally once daily (QD) for 12 weeks.
  Interventions: Drug: DC-806
- DC-806 800 mg BID (Experimental): Participants received 800 mg of DC-806 tablets orally twice daily for 12 weeks.
  Interventions: Drug: DC-806

INTERVENTIONS:
Drug: DC-806 — DC-806 was supplied as tablets to be administered orally.
  Arms: DC-806 200 mg BID; DC-806 400 mg BID; DC-806 600 mg QD; DC-806 800 mg BID
Other: Placebo — Matching placebo was supplied as tablets to be administered orally.
  Arms: Placebo

SUMMARY:
This was a 12-week treatment, multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-ranging study to evaluate the efficacy and safety of DC-806 in participants with moderate to severe plaque psoriasis. This study evaluated the efficacy, safety, tolerability, and pharmacokinetics (PK) of multiple oral doses of DC-806 in participants with moderate to severe plaque psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, 18 to 70 years of age
* Body mass index (BMI) of 18 to 40 kg/m2
* All of the following psoriasis criteria:

  * Clinical diagnosis of plaque psoriasis for ≥6 months before the Baseline visit
  * Stable moderate to severe chronic plaque psoriasis, defined as ≥10% BSA psoriasis involvement, sPGA score of ≥3, and PASI score ≥12 at the Screening and Baseline visits
  * Candidate for phototherapy or systemic therapy, as assessed by the Investigator
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must be willing to use a highly effective method of contraception during the study and for ≥30 days after the last dose of study drug
* Willing to discontinue topical and/or systemic therapies for psoriasis before the first dose of study drug

Key Exclusion Criteria:

* Have had a clinically significant flare of psoriasis during the 12 weeks before the Baseline visit, as assessed by the Investigator
* History of erythrodermic psoriasis, generalized or localized pustular psoriasis, predominantly guttate psoriasis, medication-induced or medication-exacerbated psoriasis
* History of chronic infections including human immunodeficiency virus (HIV) or viral hepatitis (hepatitis B virus [HBV], hepatitis C virus [HCV])
* History of active tuberculosis (TB)
* History or evidence of active infection (including but not limited to coronavirus disease 2019 [COVID-19] infection) and/or febrile illness within 7 days, serious infections leading to hospitalization and intravenous antibiotic treatment within 90 days, or serious infection requiring antibiotic treatment within 30 days before the first dose of study drug
* History of malignancy or lymphoproliferative disease except resected cutaneous squamous cell or basal cell carcinoma that has been treated without recurrence
* Presence of active suicidal ideation, or positive suicide behavior using the "Baseline/Screening" version of the Columbia Suicide Severity Rating Scale (C-SSRS) and with either of the following criteria:

  * History of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt) within 5 years before the Screening visit
  * Suicidal ideation in the past month before the Screening visit as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Baseline/Screening" version of the C-SSRS
* Participant has experienced primary failure (no response at approved doses after ≥3 months of therapy) to one or more therapeutic agents targeted to IL-17 (including but not limited to secukinumab, ixekizumab, brodalumab, bimekizumab)
* Systemic use of known strong and moderate cytochrome P450 (CYP)3A4 inhibitors or strong CYP3A4 inducers from Screening through the end of the study
* A 12-lead electrocardiogram (ECG) at Screening that demonstrates clinically significant abnormalities or criteria associated with QT interval abnormalities including prolongation of QT interval corrected for heart rate using Fridericia's formula (QTcF) (>500 msec)
* Laboratory values meeting the following criteria within the screening period before the first dose of study drug:

  * Serum aspartate transaminase ≥2× upper limit of normal (ULN)
  * Serum alanine transaminase ≥2×ULN
  * Serum total, direct, or indirect bilirubin ≥2.0 mg/dL; except for participants with isolated elevation of indirect bilirubin relating to a confirmed diagnosis of Gilbert syndrome
  * Estimated glomerular filtration rate (GFR) by simplified 4-variable Modification of Diet in Renal Disease (MDRD) formula <45 mL/min/1.73m2
  * Total white blood cell count <3000/μL
  * Absolute neutrophil count <1500/μL
  * Platelet count <100,000/μL
  * Hemoglobin <9 g/dL
* In the opinion of the Investigator or Sponsor, have any uncontrolled clinically significant laboratory abnormality that would affect interpretation of study data or the participant's enrollment in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (56):
- United States (13):
  - First OC Dermatology, Fountain Valley, California
  - Clinical Science Institute, Santa Monica, California
  - Driven Research LLC, Coral Gables, Florida
  - Kirsch Dermatology - Probity - PPDS, Naples, Florida
  - GCP Global Clinical Professionals, LLC, St. Petersburg, Florida
  - ForCare Clinical Research - CenExel FCR - PPDS, Tampa, Florida
  - The Indiana Clinical Trials Center, PC, Plainfield, Indiana
  - Dermatology Specialists Research - 501 S 2nd St, Louisville, Kentucky
  - DICE Therapeutics Study Site, New York, New York
  - Dermatologists of Southwest Ohio - Probity - PPDS, Mason, Ohio
  - Paddington Testing Company Inc, Philadelphia, Pennsylvania
  - Center for Clinical Studies - Webster, Webster, Texas
  - Virginia Clinical Research Inc, Norfolk, Virginia
- Canada (11):
  - Alberta DermaSurgery Centre - Probity - PPDS, Edmonton, Alberta
  - Enverus Medical Research - Probity - PPDS, Surrey, British Columbia
  - Wiseman Dermatology Research Inc. - Probity - PPDS, Winnipeg, Manitoba
  - CCA Medical Research - Probity - PPDS, Ajax, Ontario
  - SimcoDerm Medical and Surgical Dermatology Centre - Probity - PPDS, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - Lynderm Research Inc. - Probity - PPDS, Markham, Ontario
  - DermEdge Research Probity - PPDS, Mississauga, Ontario
  - DICE Therapeutics Study Site, North York, Ontario
  - Alliance Clinical Trials - Probity - PPDS, Waterloo, Ontario
  - Centre de Recherche Dermatologique du Quebec metropolitain (CRDQ), Québec
- Czechia (4):
  - Fakultni nemocnice Kralovske Vinohrady - CRC - PPDS, Prague, Praha, Hlavní Mesto
  - CCR Prague s.r.o. - PRATIA - PPDS, Prague, Praha, Hlavní Mesto
  - CCR Prague s.r.o. - PRATIA - PPDS, Prague
  - DICE Therapeutics Study Site, Prague
- Germany (9):
  - DICE Therapeutics Study Site, Erlangen, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - DICE Therapeutics Study Site, Bonn, North Rhine-Westphalia
  - DICE Therapeutics Study Site, Münster, North Rhine-Westphalia
  - DICE Therapeutics Study Site, Leipzig, Saxony
  - DICE Therapeutics Study Site, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - DICE Therapeutics Study Site, Lübeck
  - DICE Therapeutics Study Site, Tübingen
- Hungary (6):
  - Allergo-Derm Bakos Kft., Szolnok, Jász-Nagykun-Szolnok
  - DICE Therapeutics Study Site, Kaposvár, Somogy County
  - DICE Therapeutics Study Site, Szombathely, Vas County
  - Semmelweis Egyetem, Budapest
  - DICE Therapeutics Study Site, Gyöngyös
  - MedMare Bt, Veszprém
- Poland (8):
  - Cityclinic Przychodnia lekarsko psychologiczna Matusiak sp.p, Wroclaw, Lower Silesian Voivodeship
  - Wro Medica, Wroclaw, Lower Silesian Voivodeship
  - Dermoklinika-Centrum Medyczne s.c, Lódz, Lódzkie
  - Centrum Medyczne Reuma Park NZOZ, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Fryderyka Chopina w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - ClinicMed Daniluk, Nowak Spólka Komandytowa, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Angelius Provita, Katowice, Silesian Voivodeship
  - Laser Clinic S.C., Szczecin, West Pomeranian Voivodeship
- Spain (3):
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - CHUS - H. Clinico U. de Santiago, Santiago de Compostela
- United Kingdom (2):
  - Synexus Merseyside Clinical Research Centre, Liverpool, Lancashire
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | DC-806 200 mg BID | DC-806 400 mg BID | DC-806 600 mg QD | DC-806 800 mg BID
Started | 44 | 45 | 46 | 47 | 47
Received at Least One Dose of the Study Drug | 44 | 44 | 46 | 47 | 47
Safety Analysis Set (All randomized participants who received at least one dose of the study drug, with participants grouped based on the treatment they actually received. If participants received multiple treatments (e.g., DC-806 and placebo), the highest dose received was considered their actual treatment.) | 43 | 44 | 46 | 48 (One participant from the placebo group mistakenly received 600 mg of DC-806 at one visit and was grouped under 'DC-806 600 mg QD.') | 47
Completed | 32 | 31 | 40 | 40 | 44
Not Completed | 12 | 14 | 6 | 7 | 3
Not completed — Withdrawal by Subject | 11 | 10 | 4 | 3 | 2
Not completed — Lost to Follow-up | 0 | 2 | 2 | 2 | 1
Not completed — Significant protocol noncompliance | 0 | 1 | 0 | 0 | 0
Not completed — Eligibility criteria not met | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor's decision | 0 | 0 | 0 | 1 | 0
Not completed — Investigator's decision | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy of his partner | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of the study drug.
Groups:
- Placebo: Participants received placebo tablets orally twice daily for 12 weeks.
- DC-806 200 mg BID: Participants received 200 mg of DC-806 tablets orally twice daily for 12 weeks.
- DC-806 600 mg QD: Participants received 600 mg of DC-806 tablets orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | DC-806 200 mg BID | DC-806 400 mg BID | DC-806 600 mg QD | DC-806 800 mg BID | Total
Number analyzed (Participants) | 44 | 44 | 46 | 47 | 47 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (14.24) | 42.3 (12.68) | 46.0 (12.35) | 41.6 (14.25) | 43.4 (13.76) | 44.0 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 14 | 14 | 17 | 72
  Male | 33 | 28 | 32 | 33 | 30 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 2 | 6 | 4 | 21
  Not Hispanic or Latino | 39 | 38 | 43 | 40 | 41 | 201
  Unknown or Not Reported | 0 | 2 | 1 | 1 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 6 | 3 | 2 | 3 | 5 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3 | 1 | 7
  White | 35 | 36 | 43 | 41 | 40 | 195
  More than one race | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving ≥75% Reduction From Baseline in Psoriasis Area and Severity Index (PASI-75) at Week 12
Description: Participants achieving a PASI-75 without the use of other background antipsoriasis therapy were considered responders. The PASI quantifies the severity of a psoriasis based on lesion severity and the percent of body surface area (BSA) affected. Erythema, thickness, and scaling are scored on a scale of 0 (none) to 4 (very severe) on 4 anatomic regions of the body: head, trunk, upper limbs, and lower limbs. Degree of involvement on each of the 4 anatomic regions is scored on a scale of 0 (no involvement) to 6 (90% to 100% involvement). The sum of severity scores for erythema, thickness, and scaling is multiplied by the degree of involvement for each anatomic region, and then multiplied by a constant corresponding to the region's percent BSA (0.1, 0.3, 0.2, and 0.4 for the above 4 regions, respectively). The resultant score for each anatomic region is then summed to yield the final PASI score. It ranges from 0 to 72, with higher scores reflecting greater disease severity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | DC-806 200 mg BID | DC-806 400 mg BID | DC-806 600 mg QD | DC-806 800 mg BID
Number analyzed (Participants) | 44 | 44 | 46 | 47 | 47
percentage of participants | 13.6 | 6.8 | 21.7 | 17 | 36.2
Statistical Analysis 1: Comparison: Placebo vs DC-806 200 mg BID; Test type: Superiority; p = 0.4839, Fisher Exact; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.07 to 2.37] — DC-806 200 mg BID compared to Placebo
Statistical Analysis 2: Comparison: Placebo vs DC-806 400 mg BID; Test type: Superiority; p = 0.4111, Fisher Exact; Odds Ratio (OR) = 1.76, 95% CI 2-sided [0.51 to 6.49] — DC-806 400 mg BID compared to Placebo
Statistical Analysis 3: Comparison: Placebo vs DC-806 600 mg QD; Test type: Superiority; p = 0.7744, Fisher Exact; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.36 to 4.99] — DC-806 600 mg QD compared to Placebo
Statistical Analysis 4: Comparison: Placebo vs DC-806 800 mg BID; Test type: Superiority; p = 0.0164, Fisher Exact; Odds Ratio (OR) = 3.59, 95% CI 2-sided [1.15 to 12.37] — DC-806 800 mg BID compared to Placebo

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and TEASs Leading to Treatment Discontinuations
Description: * A TEAE was defined as any adverse event that began on or after the first dose of study drug or began before the first dose of study drug and worsened on or after the first dose of study drug.
  * An SAE is any untoward medical occurrence that results in 1 of the following: death, initial or prolonged inpatient hospitalization, a life-threatening experience (that is, immediate risk of dying), persistent or significant disability/incapacity, congenital anomaly/birth defect, or important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require intervention to prevent 1 of the other outcomes listed in the definition above.
Time Frame: Baseline through End of follow-up (Up to 16 weeks)
Population: All participants from the safety analyses set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DC-806 200 mg BID | DC-806 400 mg BID | DC-806 600 mg QD | DC-806 800 mg BID
Number analyzed (Participants) | 43 | 44 | 46 | 48 | 47
Participants
  TEAEs | 12 | 19 | 20 | 22 | 27
  SAEs | 0 | 0 | 0 | 0 | 1
  TEASs leading to treatment discontinuations | 1 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline through End of follow-up (Up to 16 weeks)
Description: All participants from the safety analyses set.
Arm/Group | Placebo | DC-806 200 mg BID | DC-806 400 mg BID | DC-806 600 mg QD | DC-806 800 mg BID
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/44 | 0/46 | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44 | 0/46 | 0/48 | 1/47
Other Adverse Events (participants affected / at risk) | 5/43 | 10/44 | 6/46 | 15/48 | 10/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | DC-806 200 mg BID (N=44) | DC-806 400 mg BID (N=46) | DC-806 600 mg QD (N=48) | DC-806 800 mg BID (N=47)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=43) | DC-806 200 mg BID (N=44) | DC-806 400 mg BID (N=46) | DC-806 600 mg QD (N=48) | DC-806 800 mg BID (N=47)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 7 (9) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 7 (8) | 5 (5) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT05896527/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT05896527/SAP_001.pdf